CLINICAL TRIAL: NCT00370266
Title: Intravitreal Triamcinolone for Acute Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8247
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: Macular edema; Branch retinal vein occlusion; Intravitreal triamcinolone; Macular thickness; Retinal neovascularization
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema; Retinal Neovascularization | interventions — Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone

SUMMARY:
The purpose of this study is to determine whether intraocular injection of triamcinolone is effective in the treatment of macular edema in acute branch retinal vein occlusion.

DETAILED DESCRIPTION:
Intravitreal triamcinolone has recently been shown to have beneficial effect on chronic macular edema due to vein occlusion and preventive effect on neovascularization. Hypothetically, prevention of macular derangement by reducing the amount of edema from early phase after occlusion until restoration of collaterals seems to be helpful in these eyes. To our knowledge, no prospective randomized clinical trial, considering both macular changes and preventive effect on neovascularization has been published for intravitreal triamcinolone in acute branch retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Eyes suffering from branch retinal vein occlusion with less than 2 months duration.

Exclusion Criteria:

* Monocularity,
* Previous intraocular surgery or laser therapy
* Glaucoma or ocular hypertension
* Significant media opacity
* Existence of traction on the macula
* Visual acuity ≥20/40
* Signs of chronicity (such as cilioretinal and/or retinal shunt vessels)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-02; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Central macular thickness

SECONDARY OUTCOMES:
Visual acuity
Retinal neovascularization
Intraocular pressure
Cataract progression

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Ramezani, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Alireza Ramezani, MD, Tehran, Tehran Province, Iran